CLINICAL TRIAL: NCT07140705
Title: A Personalized Virtual Reality Experience for Promoting Well-Being and Psychological Flexibility in General Practitioners: a Feasibility Study
Brief Title: Personalized Virtual Reality for Promoting Well-Being and Psychological Flexibility in General Practitioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Italian Ministry of University and Research (MUR) (Unknown); European Union (Other)
Responsible Party: Principal Investigator, Daniela Villani, Associate Professor in General Psychology, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19/25
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Virtual reality; Transformative Experience; Acceptance and Commitment Therapy; General Practitioners; Personal values; Committed action; Psychological flexibility
MeSH Terms: interventions — General Practitioners

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Other: Transformative Virtual Reality Experience and ACT for General Practitioners

INTERVENTIONS:
Other: Transformative Virtual Reality Experience and ACT for General Practitioners — This intervention consists of an individual, in-person session in which each participant engages in a 10-minute transformative Virtual Reality (VR) experience entitled "The River and the Leaf", delivered through the Meta Quest 3 headset. Drawing on Acceptance and Commitment Therapy (ACT) metaphors, participants are guided to reflect on key aspects of the experience, their professional challenges, and the personal resources available to them. Following the VR session, participants are supported in clarifying the values that guide their everyday actions. After the in-person session, all participants are encouraged to identify and implement committed actions aligned with their values over the subsequent two weeks, supported by two dedicated audio tracks.

SUMMARY:
General Practitioners (GPs) face significant daily challenges, and promoting their well-being is essential. In particular, psychological flexibility (PF) is a key indicator of well-being. PF, conceptualized within Acceptance and Commitment Therapy (ACT), supports adaptation to change and fosters adaptive responses to demanding and complex situations. ACT identifies six core processes, which can be grouped into two functional units: the mindful acceptance of one's thoughts and emotions (acceptance, cognitive defusion, openness to internal experiences), and the commitment to engaging in actions that enrich one's life (values and committed action).

This project will investigate the feasibility of a transformative metaphorical Virtual Reality (VR) experience to promote psychological flexibility and well-being in GPs. Specifically, this goal will be pursued through the integration of a metaphorical virtual experience, previously validated by the research team for its capacity to foster a transformative experience (TE)-that is, an experience that enables individuals to explore new ways of thinking and contributes to reshaping self-perception-with guided reflection on personal values and support in enacting value-consistent behaviors.

A total of 25 GPs will participate in a single in-person session involving a 10-minute transformative VR experience ("The River and the Leaf"). Drawing on ACT metaphors, participants will be guided to reflect on aspects of the experience, on the professional challenges they face, and on the personal resources available to them. Following this experience, they will be supported in identifying the values that guide their everyday actions. After the in-person session, all participants will be encouraged to identify and implement value-based committed actions over the following two weeks, supported by two audio tracks.

ELIGIBILITY:
Inclusion Criteria:

* being a General Practitioner and having an adequate understanding of the Italian language.

Exclusion Criteria:

* having pre-existing medical conditions that prevent the use of the Meta Quest 3 headset:
* presence of binocular visual abnormalities;
* history of seizures or epileptic conditions;
* presence of cardiac pacemakers, defibrillators, or implanted devices;
* use of hearing aids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
The Comprehensive assessment of ACT (CompACT) | This questionnaire will be administered at T0 (baseline) and at T2 (post-intervention, i.e., two weeks after the individual in-person session).
  This self-report scale was developed by Francis et al. (2016; Giovannetti et al., 2022) to measure psychological flexibility. The scale consists of 23 items, which can be answered using a 6-point Likert scale, where 0 indicates "completely disagree" and 6 "completely agree." The questionnaire is divided into three subscales: Openness to Experience (OE), Behavioral Awareness (BA), and Valued Action (VA), which correspond to the three pillars of psychological flexibility. Higher scores on the CompACT indicate greater psychological flexibility.
Mental Health Continuum Short Form (MHC-SF) | This questionnaire will be administered at T0 (baseline) and at T2 (post-intervention, i.e., two weeks after the individual in-person session).
  This self-report scale was developed by Keyes (2002; Petrillo et al., 2015) to measure emotional, social, and psychological well-being. The scale consists of 14 items, which can be answered using a 6-point Likert scale, where 0 indicates "never" and 5 "every day." To assess the three dimensions, the questionnaire is divided into three subscales: the Emotional Well-Being scale (EWB, items 1-3), the Social Well-Being scale (SWB, items 4-8), and the Psychological Well-Being scale (PWB, items 9-14). Higher scores on the MHC-SF indicate greater well-being.
Visual Analogue Scale (VAS) for the assessment of emotions | This questionnaire will be administered at T0 (baseline) and at T1 (immediately after the VR experience).
  This scale aims to measure the intensity of positive and negative emotions (joy, contentment, pride, love, compassion, awe, hope, gratitude, sadness, fear, anger, admiration, inspiration, and awe) (Shiota et al., 2006; Cloos et al., 2023). The intensity can be expressed using a Likert scale, where 0 corresponds to "not at all" and 10 to "very much."
Ad hoc questionnaire to investigate the impact of the VR transformative experience | This questionnaire will be administered at T1 (immediately after the VR experience).
  This 6-item questionnaire is designed to evaluate the transformative experience, its pleasantness, and its impact on self-expansion. Responses are provided on a 7-point Likert scale, where 1 indicates "not at all" and 7 indicates "very much."

SECONDARY OUTCOMES:
Slater Usoh Steed Presence Questionnaire (SUS) | This questionnaire will be administered at T1 (immediately after the VR experience).
  This self-report scale was developed by Usoh et al. (2000) to assess the user's sense of presence in the virtual environment. The instrument consists of 6 items, which are rated on a 7-point Likert scale. Higher scores on the SUS indicate a greater sense of presence.
Valued Living Questionnaire (VLQ) | This questionnaire will be administered at T1 (after the VR experience) and at T2 (post-intervention, i.e., two weeks after the individual in-person session).
  This questionnaire is designed to assess valued living and is divided into two sections (Wilson et al., 2002; Miselli et al., 2008). In the first section, participants are asked to rate the importance of 10 life domains on a 10-point Likert scale (where 1 = not at all important and 10 = extremely important). The life domains are: (1) family, (2) marriage/partnership/intimate relationships, (3) parenting, (4) friendship, (5) work, (6) education, (7) recreation, (8) spirituality, (9) citizenship, and (10) self-care. The second section asks participants to rate the extent to which their actions over the past week were consistent with each value/domain. Responses are given on a 10-point Likert scale (where 1 = not at all consistent and 10 = extremely consistent).
Maslach Burnout Inventory (MBI) | This questionnaire will be administered at T0 (baseline) and at T2 (post-intervention, i.e., two weeks after the individual in-person session).
  This questionnaire was developed by Maslach et al. (1997) to measure levels of burnout. It consists of 16 items rated on a 7-point Likert scale, where 0 corresponds to "never" and 6 to "every day." The questionnaire is divided into three subscales: Emotional Exhaustion (EE), Depersonalization (DP), and Reduced Personal Accomplishment (PA), which represent the three core dimensions of burnout.

CONTACTS AND LOCATIONS:
Locations (1):
- Università Cattolica del Sacro Cuore, Milan, Milano, Italy